CLINICAL TRIAL: NCT02528539
Title: Prevention of Secondary Lymphedema by Utilizing Self-management Education in Conjunction With Acupuncture Among Breast Cancer Patients Who Are at High Risk of Developing Lymphedema
Brief Title: Prevention of Lymphedema Among Breast Cancer Patients Through Implementation of an Integrative Therapy Program (ITP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huntington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Suzie Kline, PhD, NP, LAc, Huntington Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HMH2015.002
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Lymphedema
Keywords: Prevention; lymphedema; acupuncture; self-management
MeSH Terms: conditions — Lymphedema | interventions — Inosine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ITP (Integrative Thearpy Program) (Experimental): This ITP intervention consists of two distinct phases, Phase I, the active treatment phase and Phase II, the follow-up phase.
  Phase I (Intervention phase) begins post-operatively in 4-6 weeks with a baseline visit that includes 30-minute acupuncture treatment, followed by the 30-minute self-management educational session, and the participants will return weekly for 10 weeks.
  Phase II (Follow up phase) begins at month 6 and ends at month 18 from the surgery. The phase II consists of 1-hour quarterly ITP therapy at months 6, 9, 12, 15, and 18 and monthly telephone visits between ITP therapies at months 7, 8, 10, 11, 13, 14, 16, and 17. Self-management reinforcement and support will be implemented during telephone follow up visits
  Interventions: Other: ITP

INTERVENTIONS:
Other: ITP — The study participants will receive weekly acupuncture treatment plus education on self-management for 10 weeks after axillary node dissection, then a total of five follow up acupuncture treatments once every 3 months at 6, 9, 12, 15, and 18 months. The education and self management will be reinforced monthly by telephone visit.
  Acupuncture points include: LI 4, LV3, HT3, SP9, GB 20, KD 3, Yintang, and Ashi points
  Other Names: Integrative Therapy Program

SUMMARY:
Introduction: Breast cancer women who are treated with axillary node dissection are at increased risk for lymphedema - the lifetime risk in these women is estimated at 15-50% and the risk can significantly increase with chemotherapy and radiation therapy

Objectives:

1. To evaluate the feasibility and effectiveness of implementing the integrative therapy program (ITP) intervention. ITP consists of self-management education in conjunction with acupuncture.
2. To determine if ITP affects quality of life, self-efficacy, lymphedema knowledge, pain, and early detection and management of lymphedema.

Design: the exploratory study aims to evaluate the feasibility and benefits of the integrative therapy program (ITP) intervention post-operatively for 18 months.

Subjects: Women with breast cancer treated with axillary node dissection with normal baseline pre-operative bioimpedance (L-dex U400) score.

Sample size: 30 subjects

DETAILED DESCRIPTION:
Recruitment and Intervention:

The study participants are recruited by their breast surgeon after they undergo axillary node dissection surgery. 4-6 weeks following surgery, the participants will receive a combination of acupuncture and self management education .

Contents of self-management education include:

1. Lymphedema knowledge: functions of the lymphatic system, anatomy of the lymph nodes and direction of the lymphatic drainage, risk factors that could precipitate lymphedema, the signs and symptoms of lymphedema and infection, and lymphedema resources.
2. Selfcare techniques:healthy diet (eating whole food encouraged), neck, shoulder and chest wall stretching exercises, walk daily, self-manual lymphatic drainage with deep breathing techniques, and self-acupressure over eighteen months following their surgery.

Outcome measurements include: L-Dex U400 measurement, arm circumference, pain scale, self-efficacy, and lymphedema knowledge, and Functional Assessment of Cancer Therapy-Breast FACT-B.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to read and understand the informed consent form and have the capacity to give consent.
2. Adults age 18 and older
3. Subject with a newly diagnosed stage I-III breast cancer with a documented pre-operative baseline L-Dex U400 who underwent axillary lymph node dissection within 4-6 weeks prior to enrollment.
4. Subjects must be able to return to the study site for the duration of the study (18 months).

Exclusion Criteria:

1. Subjects who do not read or understand the informed consent are ineligible.
2. Subjects who have any contraindications to the affected upper-limb exercises, which include congestive heart failure, cardiac arrhythmia, deep vein thrombosis, infectious disease complications such as cellulitis and lymphangitis.
3. Women with double mastectomy with axillary node dissection bilaterally.
4. Women with a prior history of axillary surgeries in the ipsilateral side and/or primary lymphedema
5. Women with metal implants (e.g. shoulder replacement) or cardiac implants (e.g. automated implanted cardiac defibrillator (AICD) or pacemaker).
6. All subjects with objective or subjective signs and symptoms of lymphedema.
7. Women of childbearing age who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Bioimpedance (L-dex U400) | 18 months
  use L-dex machine
Arm circumference measurements of the upper limbs using at 4 cm interval | 18 months
  measure the circumference in centimeters

SECONDARY OUTCOMES:
Self-Efficacy Scale | 18 months
  questionnaires
Lymphedema Knowledge Scale | 18 months
  questionnaires
Quality of Life (Functional Assessment of Cancer Therapy-Breast) | 18 months
  survey
Wong-Baker FACES Pain Scale | 18 months
  1-10 scale

CONTACTS AND LOCATIONS:
Overall Officials: Suzie S Kline, PhD, Principal Investigator — Huntington Hospital
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armer JM, Brooks CW, Stewart BR. Limitations of self-care in reducing the risk of lymphedema: supportive-educative systems. Nurs Sci Q. 2011 Jan;24(1):57-63. doi: 10.1177/0894318410389058. PMID 21220577
- [Background] Armer JM, Shook RP, Schneider MK, Brooks CW, Peterson J, Stewart BR. Enhancing Supportive-Educative Nursing Systems to Reduce Risk of Post-Breast Cancer Lymphedema. Self Care Depend Care Nurs. 2009 Oct;17(1):6-15. PMID 22872189
- [Background] Beaulac SM, McNair LA, Scott TE, LaMorte WW, Kavanah MT. Lymphedema and quality of life in survivors of early-stage breast cancer. Arch Surg. 2002 Nov;137(11):1253-7. doi: 10.1001/archsurg.137.11.1253. PMID 12413312
- [Background] Binkley JM, Harris SR, Levangie PK, Pearl M, Guglielmino J, Kraus V, Rowden D. Patient perspectives on breast cancer treatment side effects and the prospective surveillance model for physical rehabilitation for women with breast cancer. Cancer. 2012 Apr 15;118(8 Suppl):2207-16. doi: 10.1002/cncr.27469. PMID 22488695
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Cassileth BR, Van Zee KJ, Chan Y, Coleton MI, Hudis CA, Cohen S, Lozada J, Vickers AJ. A safety and efficacy pilot study of acupuncture for the treatment of chronic lymphoedema. Acupunct Med. 2011 Sep;29(3):170-2. doi: 10.1136/aim.2011.004069. Epub 2011 Jun 18. PMID 21685498
- [Background] Cemal Y, Pusic A, Mehrara BJ. Preventative measures for lymphedema: separating fact from fiction. J Am Coll Surg. 2011 Oct;213(4):543-51. doi: 10.1016/j.jamcollsurg.2011.07.001. Epub 2011 Jul 28. No abstract available. PMID 21802319
- [Background] Chang CJ, Cormier JN. Lymphedema interventions: exercise, surgery, and compression devices. Semin Oncol Nurs. 2013 Feb;29(1):28-40. doi: 10.1016/j.soncn.2012.11.005. PMID 23375064
- [Background] de Valois BA, Young TE, Melsome E. Assessing the feasibility of using acupuncture and moxibustion to improve quality of life for cancer survivors with upper body lymphoedema. Eur J Oncol Nurs. 2012 Jul;16(3):301-9. doi: 10.1016/j.ejon.2011.07.005. Epub 2011 Sep 13. PMID 21917515
- [Background] Dibble SL, Chapman J, Mack KA, Shih AS. Acupressure for nausea: results of a pilot study. Oncol Nurs Forum. 2000 Jan-Feb;27(1):41-7. PMID 10660922
- [Background] DiSipio T, Rye S, Newman B, Hayes S. Incidence of unilateral arm lymphoedema after breast cancer: a systematic review and meta-analysis. Lancet Oncol. 2013 May;14(6):500-15. doi: 10.1016/S1470-2045(13)70076-7. Epub 2013 Mar 27. PMID 23540561
- [Background] Dobos GJ, Kirschbaum B, Choi KE. The Western model of integrative oncology: the contribution of Chinese medicine. Chin J Integr Med. 2012 Sep;18(9):643-51. doi: 10.1007/s11655-012-1200-1. Epub 2012 Aug 31. PMID 22936317
- [Background] Yen TW, Fan X, Sparapani R, Laud PW, Walker AP, Nattinger AB. A contemporary, population-based study of lymphedema risk factors in older women with breast cancer. Ann Surg Oncol. 2009 Apr;16(4):979-88. doi: 10.1245/s10434-009-0347-2. Epub 2009 Feb 5. PMID 19194754
- [Background] Zimmermann A, Wozniewski M, Szklarska A, Lipowicz A, Szuba A. Efficacy of manual lymphatic drainage in preventing secondary lymphedema after breast cancer surgery. Lymphology. 2012 Sep;45(3):103-12. PMID 23342930
- [Background] Stout Gergich NL, Pfalzer LA, McGarvey C, Springer B, Gerber LH, Soballe P. Preoperative assessment enables the early diagnosis and successful treatment of lymphedema. Cancer. 2008 Jun 15;112(12):2809-19. doi: 10.1002/cncr.23494. PMID 18428212
- [Background] Rottmann N, Dalton SO, Christensen J, Frederiksen K, Johansen C. Self-efficacy, adjustment style and well-being in breast cancer patients: a longitudinal study. Qual Life Res. 2010 Aug;19(6):827-36. doi: 10.1007/s11136-010-9653-1. Epub 2010 Apr 17. PMID 20401551
- [Background] Meng Z, Garcia MK, Hu C, Chiang J, Chambers M, Rosenthal DI, Peng H, Zhang Y, Zhao Q, Zhao G, Liu L, Spelman A, Palmer JL, Wei Q, Cohen L. Randomized controlled trial of acupuncture for prevention of radiation-induced xerostomia among patients with nasopharyngeal carcinoma. Cancer. 2012 Jul 1;118(13):3337-44. doi: 10.1002/cncr.26550. Epub 2011 Nov 9. PMID 22072272
- [Background] Mansel RE, Fallowfield L, Kissin M, Goyal A, Newcombe RG, Dixon JM, Yiangou C, Horgan K, Bundred N, Monypenny I, England D, Sibbering M, Abdullah TI, Barr L, Chetty U, Sinnett DH, Fleissig A, Clarke D, Ell PJ. Randomized multicenter trial of sentinel node biopsy versus standard axillary treatment in operable breast cancer: the ALMANAC Trial. J Natl Cancer Inst. 2006 May 3;98(9):599-609. doi: 10.1093/jnci/djj158. PMID 16670385
- [Background] MacPherson H, Thomas K, Walters S, Fitter M. A prospective survey of adverse events and treatment reactions following 34,000 consultations with professional acupuncturists. Acupunct Med. 2001 Dec;19(2):93-102. doi: 10.1136/aim.19.2.93. PMID 11829165
- [Background] Langer I, Guller U, Berclaz G, Koechli OR, Schaer G, Fehr MK, Hess T, Oertli D, Bronz L, Schnarwyler B, Wight E, Uehlinger U, Infanger E, Burger D, Zuber M. Morbidity of sentinel lymph node biopsy (SLN) alone versus SLN and completion axillary lymph node dissection after breast cancer surgery: a prospective Swiss multicenter study on 659 patients. Ann Surg. 2007 Mar;245(3):452-61. doi: 10.1097/01.sla.0000245472.47748.ec. PMID 17435553
- [Background] Hibbard JH, Greene J, Overton V. Patients with lower activation associated with higher costs; delivery systems should know their patients' 'scores'. Health Aff (Millwood). 2013 Feb;32(2):216-22. doi: 10.1377/hlthaff.2012.1064. PMID 23381513
- [Background] Vicini FA, Kestin L, Chen P, Benitez P, Goldstein NS, Martinez A. Limited-field radiation therapy in the management of early-stage breast cancer. J Natl Cancer Inst. 2003 Aug 20;95(16):1205-10. doi: 10.1093/jnci/djg023. PMID 12928345
- [Background] Erickson VS, Pearson ML, Ganz PA, Adams J, Kahn KL. Arm edema in breast cancer patients. J Natl Cancer Inst. 2001 Jan 17;93(2):96-111. doi: 10.1093/jnci/93.2.96. PMID 11208879
- [Background] Easom LR. Concepts in health promotion. Perceived self-efficacy and barriers in older adults. J Gerontol Nurs. 2003 May;29(5):11-9. doi: 10.3928/0098-9134-20030501-05. PMID 12765007